CLINICAL TRIAL: NCT05234268
Title: Comparative Effectiveness of Manual Cervical Traction, Passive Accessory Intervertebral Movements and Active Strength Training in the Management of Cervical Radiculopathy
Brief Title: Cervical Traction, Passive Accessory Intervertebral Movements and Active Strength Training in Cervical Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01060 Yusra Arif
Record Dates: First submitted 2022-02-01; First posted 2022-02-10 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Cervical Radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Manual Cervical Traction (Experimental): The patient is in supine lying. The head and neck of patient are held in the hands of the practitioner, and then a gentle traction of a pulling force is applied. Intermittent periods of traction can be applied, holding each position for about 10 seconds. Traction is usually applied at about 20-30 degrees of neck flexion.
  Interventions: Other: Manual Cervical Traction
- Passive Accessory Intervertebral Movements (Experimental): Patient lying in prone. Therapist stands to side of patient placing their pisiform/ulnar surface of hand over the selected spinous process (SP) with their wrist in full extension. Other hand placed on top of hand to reinforce. Therapist's shoulders should be directly above the SP with elbows slightly bent. Therapist uses their body weight to apply a PA force to the selected SP by leaning their body over their arms and performing rocking movements to provide oscillatory movements of the vertebra.
  Interventions: Other: Passive Accessory Intervertebral Movements
- Active Strength Training (Experimental): The progression of exercises will be done using different colours of Thera-band indicating varied resistance
  Interventions: Other: Active Strength Training

INTERVENTIONS:
Other: Manual Cervical Traction — Time: 20 minutes Duration: thrice a week for 4 weeks.
  Position:
  The patient is in supine lying. The head and neck of patient are held in the hands of the practitioner, and then a gentle traction of a pulling force is applied. Intermittent periods of traction can be applied, holding each position for about 10 seconds. Traction is usually applied at about 20-30 degrees of neck flexion.
  Arms: Manual Cervical Traction
Other: Passive Accessory Intervertebral Movements — Time: 20 minutes Duration: thrice a week for 4 weeks
  Position:
  Patient lying in prone. Therapist stands to side of patient placing their pisiform/ulnar surface of hand over the selected spinous process (SP) with their wrist in full extension.
  Other hand placed on top of hand to reinforce. Therapist's shoulders should be directly above the SP with elbows slightly bent. Therapist uses their body weight to apply a PA force to the selected SP by leaning their body over their arms and performing rocking movements to provide oscillatory movements of the vertebra.
  Arms: Passive Accessory Intervertebral Movements
Other: Active Strength Training — Time: 20 minutes Duration: thrice a week for 4 weeks. The progression of exercises will be done using different colors of Thera-band indicating varied resistance. (A) Resistive lateral flexion of uninvolved side.
  Position:
  The patient is in sitting position. By the help of thera-band patient will actively flex the neck against resistance on the uninvolved side.
  Arms: Active Strength Training

SUMMARY:
To determine the effectiveness of Manual Cervical Traction, Passive Accessory Intervertebral Movements (PAIVMs) and Active strength training in the management of cervical radiculopathy. To compare the effectiveness of Manual Cervical Traction, Passive Accessory Intervertebral Movements (PAIVMs) and Active strength training in the management of cervical radiculopathy.

DETAILED DESCRIPTION:
Cervical radiculopathy is a clinical condition resulting from compression of cervical nerve roots near the spinal cord. Some factors that may increase the risk for developing cervical radiculopathy include age. The risk for cervical radiculopathy tends to increase with age. This study is based on three interventions (Manual Cervical traction, Passive Accessory Intervertebral Movements (PAIVMs) and Active Strength Training) individually on three separate but equal groups of participants. It will determine the most effective intervention and which intervention is superior to the other for treating cervical radiculopathy and to assist future practitioners and researchers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cervical radiculopathy due to muscle tightness or spasm (Diagnosed by Spurling's Test)
* Having complaint more than 2 months

Exclusion Criteria:

* Past history of cervical surgery
* Past history of cervical trauma
* Any inflammatory disease
* Tumor or Carcinoma
* Disco genic/ disc herniation or stenosis cause of radiculopathy.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
Pain Relief by Visual Analogue Scale (VAS) | 4 weeks
  A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms. The simplest VAS is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptom, pain, health) orientated from the left (worst) to the right (best).
Activities of daily living by Neck Disability Index (NDI) | 4 Weeks
  This questionnaire has been designed to give us information as to how your neck pain has affected your ability to manage in everyday life. Patient-completed, condition- specific, functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation.
  Each section is scored on a 0 to 5 rating scale, in which zero means "no pain" and 5 means "Worst imaginable pain".
Cervical Compression Test by Spurling's Test | 4 Weeks
  The Spurling's test (also known as Maximal Cervical Compression Test and Foraminal Compression Test) is used during a musculoskeletal assessment of the cervical spine when looking for cervical nerve root compression causing Cervical Radiculopathy. There are different ways described in the literature to perform the Spurling's test. The version that provoked upper limb symptoms the best was with the neck in extension, lateral flexion and axial compression.

SECONDARY OUTCOMES:
Cervical Range of motion by Goniometer | 4 Weeks
  A goniometer is an instrument which measures the available range of motion at a joint. Goniometer have different types; the most use is the universal standard goniometer, which is either made with plastic or metal tool. It consists of a stationary arm, a movable arm and a fulcrum.
Endurance of the deep flexors of the cervical spine by Cranio-cervical Flexion Test | 4 week
  The Craniocervical flexion test (CCFT) is a clinical test of neuromotor control including the activation and endurance of the deep flexors of the cervical spine. This test involves the subject performing a "yes" like nod which is the anatomical action of the Deep Cervical flexors, against a pressure biofeedback. The CCFT tests the neuromuscular control of the control of the deep cervical flexor muscles, the longus capitis, and colli. The test also assesses endurance of the deep cervical flexors and interaction of the deep cervical flexor muscles with the superficial flexors, i.e. the Sternocleidomastoid and the anterior scalene muscles. It can also be used as a clinical indicator of impaired activation of the deep cervical flexor muscles, to measure the muscle activity of the deep and superficial cervical muscles.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Khalid, MSPT-OMPT, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Quaid-e-Azam International Hospital, Rawalpindi, Punjab Province
  - Pakistan Railway General Hospital, Rawalpindi, Punjab Province

IPD SHARING:
Plan to Share IPD: No